CLINICAL TRIAL: NCT01108302
Title: Assessing the Effectiveness, Safety and Feasibility of Expanding Use of Oxytocin in Uniject™ by Auxiliary Nurse Midwives to Prevent Postpartum Hemorrhage: A Community-based Cluster Randomized Trial in Bagalkot, India
Brief Title: Effectiveness, Safety and Feasibility of Auxiliary Nurse Midwives' (ANM) Use of Oxytocin in Uniject™ to Prevent Postpartum Hemorrhage in India
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PATH withdrew IRB approval
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Jawaharlal Nehru Medical College Women's and Children's Health Research Unit (Unknown); PATH (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Cynthia Stanton, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAT.1429-07882-2
Record Dates: First submitted 2010-04-02; First posted 2010-04-21 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-12

CONDITIONS: Postpartum Hemorrhage
Keywords: uterotonic; oxytocin; randomized trial; India; community; hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPH Treatment only (No Intervention): Auxilliary nurse midwives will be able to treat for PPH only, not provide Oxytocin in Uniject
- Oxytocin in Uniject (Experimental): Auxilliary Nurse Midwives will provide 10IU Oxytocin in Uniject device IM immediately after delivery
  Interventions: Other: Oxytocin in Uniject

INTERVENTIONS:
Other: Oxytocin in Uniject — 10 IU Oxytocin delivered intramuscularly immediately after delivery of the baby
  Other Names: Pitocin, Syntocinon
  Arms: Oxytocin in Uniject

SUMMARY:
This cluster randomized community-based trial is designed to test the hypothesis that the intramuscular administration of 10 IU of oxytocin in Uniject™ during the third stage of labor by an Auxiliary Nurse Midwife (ANM) at births occurring in homes, Sub-Centers and Primary Health Centers in Bagalkot, India will reduce the risk of postpartum hemorrhage by 44% (from 9% to 5%) relative to home births attended by the same type of provider who does not provide the intervention drug. The study will also document correct use of oxytocin in Uniject, adverse maternal and fetal events associated with inappropriate use and a number of indicators reflecting the programmatic feasibility of implementing this intervention.

ELIGIBILITY:
Inclusion Criteria:

* gestational age >=28 wks at enrollment
* anticipate spontaneous vaginal delivery
* hemoglobin >=8 gm/dl
* delivery at home, sub-center, or primary health center
* delivery attended by Auxilliary Nurse Midwife

Exclusion Criteria:

* previous caesarean-section
* scheduled for caesarean-section
* antepartum bleeding during current pregnancy
* blood pressure >140mm of Hg systolic and >90mm of Hg diastolic
* in active labor at time of recruitment
* high risk medical conditions (diabetes, cardiac ailments, seizures, placenta previa, anticipated breech delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
postpartum hemorrhage | after delivery of baby
  blood loss >=500 ml after delivery of the baby, as measured through a plastic calibrated drape.

SECONDARY OUTCOMES:
Oxytocin use before delivery | labor and delivery
  the proportion of deliveries where oxytocin in uniject was administered prior to the delivery of the baby
stillbirth | pregnancy
  stillbirth is defined as death of a fetus after 28 weeks of gestation and before birth of the baby
neonatal death | first month of life
  neonatal death is defined as death of a live born infant prior to completion of 28 days
need for neonatal resuscitation | 0-6 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stanton, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Shivaprasad Goudar, MD, Principal Investigator — JN Medical College, Belgaum, India
Locations (1):
- Jawaharlal Nehru Medical College Women's and Children's Health Research Unit, Belagavi, Karnataka, India